CLINICAL TRIAL: NCT04615182
Title: The Portable Organ Care System (OCS™) Heart For Resuscitation, Preservation and Assessment of Hearts From Donors After Circulatory Death Continued Access Protocol (OCS DCD Heart CAP)
Brief Title: Donor After Circulatory Death Heart CAP Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TransMedics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OCS-CAR-08242020
Record Dates: First submitted 2020-10-28; First posted 2020-11-04 (Actual); Results first posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2022-09

CONDITIONS: Heart Transplant
MeSH Terms: interventions — Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- OCS Preservation (Experimental)
  Interventions: Device: Transplant

INTERVENTIONS:
Device: Transplant — To enable continued clinical access to DCD heart transplantation in the U.S. and to continue to collect additional data on the performance of the OCS Heart System to resuscitate, preserve and assess hearts donated after circulatory death for transplantation to increase the pool of donor hearts available for transplantation.

SUMMARY:
The Portable Organ Care System (OCS™) Heart for Resuscitating, Preserving and Assessing Hearts Donated after Circulatory Death Continued Access Protocol (OCS DCD Heart CAP)

DETAILED DESCRIPTION:
To enable continued clinical access to DCD heart transplantation in the U.S. and to continue to collect additional data on the performance of the OCS Heart System to resuscitate, preserve and assess hearts donated after circulatory death for transplantation to increase the pool of donor hearts available for transplantation.

ELIGIBILITY:
Recipient Inclusion Criteria:

* • Primary heart transplant candidates

  * Age ≥ 18 years old
  * Signed: (1) written informed consent document; (2) authorization to use and disclose protected health information; and (3) consent to TransMedics' use of recipients' UNOS/OPTN data and recipients' INTERMACS data.

Recipient Exclusion Criteria:

* Prior solid organ or bone marrow transplant

  * Chronic use of hemodialysis or diagnosis of chronic renal insufficiency
  * Multi-organ transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2020-11-25 (Actual); Primary Completion 2021-12-21 (Actual); Study Completion 2022-06-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (25):
- United States (25):
  - University of California San Diago, La Jolla, California
  - Cedars Sinai, Los Angeles, California
  - Stanford University, Palo Alto, California
  - Yale New Haven Hospital, New Haven, Connecticut
  - Mayo Clinic Florida, Jacksonville, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Tampa General Hospital, Tampa, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Northwestern University, Evanston, Illinois
  - St. Vincent Cardiovascular Research Institute, Indianapolis, Indiana
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Minneapolis Heart Institute, Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Nyph/Cumc, New York, New York
  - Montefiore, The Bronx, New York
  - Westchester Medical Center, Valhalla, New York
  - Duke University, Durham, North Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Sentara, Norfolk, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - University of Wisconsin, Madison, Wisconsin
  - Froedtert & the Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | OCS Preservation
Started | 90
Per Protocol Population | 83
Completed | 75
Not Completed | 15
Not completed — Re-transplanted | 2
Not completed — Protocol Violation | 6
Not completed — Death | 6
Not completed — Death and protocol violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | OCS Preservation
Number analyzed (Participants) | 83
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.1 (12.923)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 65
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 74
  Unknown or Not Reported | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 16
  White | 61
  More than one race | 0
  Unknown or Not Reported | 4

OUTCOME MEASURES:

1. Primary Outcome: Patient Survival
Description: Patient survival at 6 months post-transplant.
Time Frame: 6 months post-transplant
Population: Per protocol population reported. Two subjects were withdrawn due to re-transplant and were excluded from the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | OCS Preservation
Number analyzed (Participants) | 81
Participants | 75

2. Secondary Outcome: Utilization Rate
Description: Utilization Rate, defined as the number of eligible DCD donor hearts that met the warm ischemic time limit per protocol and were instrumented on the OCS Heart System that meet the acceptance criteria for transplantation after OCS Heart preservation divided by the total number of eligible DCD donor hearts that met the warm ischemic time limit above and were instrumented on the OCS Heart System.
Time Frame: 24 hours post transplant
Population: 95 eligible DCD donor hearts met the warm ischemic time limit per protocol and were instrumented on the OCS Heart System.
Measure: Count of Units; unit: Hearts Instrumented
Units Other Than Participants: Hearts Instrumented
Arm/Group | OCS Preservation
Number analyzed (Participants) | 83
Number analyzed (Hearts Instrumented) | 95
Hearts Instrumented | 83

ADVERSE EVENTS:
Time Frame: Serious adverse events will be collected only through Day 30 post-transplant. All-cause mortality was evaluated through 6-months post-transplant.
Description: Per the protocol, only serious adverse events (SAEs) and Heart Graft-Related SAE's (HGRSAEs) were captured in this study.
  Other [Not Including Serious] Adverse Events were not monitored/assessed, and therefore are not reported.
Arm/Group | OCS Preservation
All-Cause Mortality (participants affected / at risk) | 7/90
Serious Adverse Events (participants affected / at risk) | 53/90
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OCS Preservation (N=90)
Blood loss anaemia (Blood and lymphatic system disorders) | 1 (1)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1)
Cardiac tamponade (Cardiac disorders) | 3 (3)
Left ventricular dysfunction (Cardiac disorders) | 21 (21)
Pericardial effusion (Cardiac disorders) | 5 (6)
Pericardial haemorrhage (Cardiac disorders) | 1 (1)
Right ventricular dysfunction (Cardiac disorders) | 2 (2)
Tricuspid valve incompetence (Cardiac disorders) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Transplant rejection (Immune system disorders) | 9 (10)
COVID-19 (Infections and infestations) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 1 (1)
Fungaemia (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Sepsis (Infections and infestations) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 1 (1)
Mental status changes postoperative (Injury, poisoning and procedural complications) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Vocal cord paralysis (Nervous system disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 10 (10)
Renal failure (Renal and urinary disorders) | 2 (2)
Renal impairment (Renal and urinary disorders) | 2 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Deep vein thrombosis (Vascular disorders) | 2 (2)
Haematoma (Vascular disorders) | 2 (2)
Haemorrhage (Vascular disorders) | 4 (4)
Peripheral ischaemia (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Site shall have right to publish results. To balance this right with TransMedics' (TM) proprietary interests, site will submit manuscripts intended for publication for TM's review at least 30 days prior to submission date. TM will complete its review within 30 days of receipt. TM may request that site delete from its manuscripts any reference to TM confidential information and site shall promptly comply with such request.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-16): https://cdn.clinicaltrials.gov/large-docs/82/NCT04615182/Prot_SAP_000.pdf